CLINICAL TRIAL: NCT02708017
Title: The Analgesic Efficacy of Ultrasound Guided Bilateral Subcostal vs. Posterior Transversus Abdominis Plane Block After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Analgesic Effect of Subcostal TAP Block
Acronym: UGS-TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, DR.Karima karam khan, Dr.Karima karam khan, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2317-ane-ERC-12
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Subcostal TAP Block for Multiport Laparoscopic Cholecystectomy
Keywords: Subcostal TAP block; Posterior TAP block; Ultrasound; Laparoscopic cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-TAP block (Active Comparator): ultrasound guided bilateral subcostal TAP block
  Interventions: Procedure: Ultrasound guided bilateral subcostal TAP block
- P-TAP block (Active Comparator): ultrasound guided bilateral Posterior TAP block
  Interventions: Procedure: Ultrasound guided bilateral posterior TAP block

INTERVENTIONS:
Procedure: Ultrasound guided bilateral subcostal TAP block — ultrasound guided bilateral subcostal TAP block was performed after induction of general anaesthesia.after all aseptic measures,abdomen was prepared with antiseptic spray,with the help of portable ultrasound machine using probe frequency of 11 Mega Hertz,ultrasound probe was positioned parallel to the costal margin near the midline,the rectus abdominis muscle was identified ,probe was gradually moved laterally and obliquely along the subcostal margin and the transversus abdominis muscle identified lying posterior to the rectus muscle.the 20Gauge,100millimeter long needle was introduced at the lateral edge of the rectus muscle ,from medial to lateral,in plane of the ultrasound beam.After confirmation of the plane with saline, 20ml of 0.375% solution of bupivacaine was injected on each side of the abdomen.
  Other Names: S-TAP Block
  Arms: S-TAP block
Procedure: Ultrasound guided bilateral posterior TAP block — ultrasound guided bilateral posterior TAP block was performed after induction of general anaesthesia.after all aseptic measures,abdomen was prepared with antiseptic spray.with the help of portable ultrasound machine using probe frequency of 11Mega Hertz,ultrasound probe was positioned transversely to the abdominal wall in the midaxillary line between the iliac crest and coastal margin,and carefully moved posteriolaterally for optimal identification of plane.the 20G,100mm long needle was introduced anteriorly and in line with the probe,from medial to lateral,and advanced until it reached the fascial plane between the internal oblique and transversus abdominis muscle.upon reaching the plane ,20ml of 0.375% solution of bupivacaine was injected on each side of the abdomen.
  Other Names: P-TAP Block
  Arms: P-TAP block

SUMMARY:
The purpose of this study was to compare the analgesic efficacy of the ultrasound guided bilateral subcostal tap block with ultrasound guided bilateral posterior tap block for postoperative analgesia after laparoscopic cholecystectomy

DETAILED DESCRIPTION:
After approval from Ethics Review Committee, patients were enrolled according to the inclusion and exclusion criteria. Informed written consent for inclusion in the study was taken and during the process,patients were explained about the NRS and other secondary objectives.

Blocks were performed under ultrasound guidance immediately after induction of anesthesia.For postoperative analgesia,patients were randomly allocated in two groups using draw/ballot method assigning patients to either of the S-TAP block group or P-TAP-block group. The patients and the staff providing postoperative care and the doctor assessing the pain after surgery were blinded to group assignment. Patients in both groups received standard of care analgesia during the post-operative period i.e., I/V Ketorolac 30mg every 8 hourly, I/V Tramadol 50mg every 8hourly and as per need basis, and I/V Paracetamol 1000mg every 6 hourly Subsequent surgical procedure was performed routinely. After completion of the surgery and emergence from anesthesia, patients were shifted to the Post Anaesthesia Care Unit, and time of arrival in recovery room was taken as 0-hour and noted. Assessment for outcome measures started in recovery room, and continued till 24 hours of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 to 60 years,American society of Anaesthesiology(ASA) class I and II, admitted electively for laparoscopic cholecystectomy

Exclusion Criteria:

* Patients with known allergies to local anesthetics, who were morbidly obese because of difficulty of ultrasound guided approaches for block or having hepato-splenomegaly or any known liver disease, and those whose laparoscopic procedure is converted to open cholecystectomy for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mean postoperative static and dynamic numeric rating scale (NRS) at 24 hours | 24 hours
  To compare the mean NRS at 0hr, 1hr, 2 hrs. 6 hrs. 12 hrs. and 24hrs. post-operatively between two groups Numeric rating scale for pain,(0=no pain, 1-3= mild pain, 4-6 moderate pain, 7-10 severe pain.)

SECONDARY OUTCOMES:
Mean opioid consumption postoperatively | 24hours
  To compare post-operative mean opioid consumption in the two groups
Nausea , vomiting and sedation score | 24 hours
  To compare mean post-operative nausea, vomiting and sedation scores between the two groups.
  Nausea score (none = 0; mild = 1(requiring no medication); moderate = 2(requiring anti-emetics); severe = 3(unresponsive to anti-emetics) Sedation score (awake and alert =0; quietly awake = 1; asleep but easily roused = 2; deep sleep =3)
Surgical outcome | 24 hours
  To compare surgical outcomes in terms of early mobilization out of bed,intake of first postoperative meal,and early discharge after 24 hours of surgery between the two groups
Patient satisfaction | 24hours
  patient satisfaction is assessed by using a questionnaire at 24hours
  1. Are you satisfied with the method of your pain relief? Yes / No
  2. Would you recommend the same method of pain relief to your family/friends? Yes / No

CONTACTS AND LOCATIONS:
Overall Officials: Karima K Khan, FCPS, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: No